CLINICAL TRIAL: NCT02632968
Title: Pinhole Surgical Technique With And Without Use Of Button Application For Treatment Of Multiple Gingival Recessions: A Comparative Controlled Randomized Clinical Trial
Brief Title: Pinhole Surgical Technique With And Without Use Of Buttons For Treatment Of Multiple Gingival Recessions: RCT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_44452
Record Dates: First submitted 2015-12-15; First posted 2015-12-17 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pinhole surgery with orthodontic buttons (Active Comparator): Pinhole surgery with orthodontic buttons The selected participants were assigned in test and control. In the test group orthodontic buttons were cemented on the bid-buccal region of the crown with dual cure GIC. After administration of LA, 2 to 3 pinhole incisions were made and a full thickness muco-periosteal tunnel was raised and collagen membrane was tucked in through the pinhole incisions. The sling sutures 5-0 mersilk were placed to hold the tunnel in an advanced location using orthodontic buttons as anchoring units. Inter-dental sutures with 6-0 mersilk were also placed for stabilization of the advanced gingival tissue.
  Interventions: Procedure: Pinhole surgery with and without buttons
- Pinhole surgery without buttons (Active Comparator): Pinhole surgery without orthodontic buttons The selected participants were assigned in test and control. In the control group, after administration of LA, 2 to 3 pinhole incisions were made and a full thickness muco-periosteal tunnel was raised and collagen membrane was tucked in through the pinhole incisions till the recession defects were covered. No sutures or orthodontic buttons were used in the control site.
  Interventions: Procedure: Pinhole surgery with and without buttons

INTERVENTIONS:
Procedure: Pinhole surgery with and without buttons

SUMMARY:
Pinhole surgical technique is a novel minimally invasive, predictable, efficient, time and cost-effective technique for treatment of multiple gingival recession. This procedure involves no releasing incision, suturing or sharp dissections. It has been shown that the greater post-operative displacement of gingival margin may cause greater root coverage. Based on this hypothesis, a split mouth randomized controlled clinical trial was planned to compare the clinical outcome of pinhole surgical technique with and without the use of orthodontic buttons and sutures in the treatment of multiple gingival recessions.

DETAILED DESCRIPTION:
To achieve multiple adjacent recession coverage and an optimal integration of the associated tissues is even more challenging and a complex endeavour in comparison to isolated gingival recessions. Treatment protocol and outcome with different surgical procedures depends on a variety of factors like recession, defect size, presence or absence of keratinized tissue adjacent to the defect, width and height of inter-dental soft tissue, depth of vestibule, presence of frenum, post-operative stabilization and final position of advanced gingival margin. The final position of the GM plays a critical role in achieving CRC. Based on this hypothesis, a split mouth clinical trial was planned to compare the clinical outcome of pinhole surgical technique with and without the use of orthodontic buttons and sutures in the treatment of multiple gingival recessions.

METHOD The aim of this split-mouth randomized controlled clinical trial was to clinically compare and evaluate the effectiveness and predictability of Pinhole surgical technique alone and its modification with orthodontic buttons and sutures in 80 sites for the treatment of multiple gingival recessions and to assess the influence of these surgical procedures on the gingival and periodontal health, in the maxillary arch for six months post surgically. Gingival recession depth (GRD), Gingival margin location post-surgery, Gingival recession width (GRW), Root coverage esthetic score (RES), Complete root coverage (CRC), Probing depth (PD), Clinical attachment level (CAL), Keratinized tissue width (KTW), Plaque index (PI), Gingival index (GI), Gingival bleeding index (GBI) will be measured at baseline, 6 weeks, 3 months and 6 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Multiple (atleast two or three) Millers class I and II or combined class I and II recession defects18 affecting adjacent teeth of the maxillary arch.
* Patients with thick gingival biotypes >0.8mm.
* Presence of adequate keratinized tissue apical to recession > 1mm.
* Age group 25-55 years.
* Patients with history of compliance to oral hygiene instructions and a full mouth plaque score of <10%.
* Patients willing to participate in the study.
* American Society of Anaesthesiologists Physical Status I or II.
* No contra-indications for periodontal surgery.
* Non-Smokers.
* Patients with esthetic concerns.

Exclusion Criteria:

* Recession defects associated with caries/demineralization, restorations, and deep abrasions (step >2mm).
* No occlusal interferences.
* Teeth with evidence of pulpal pathology.
* Patients who have undergone any previous periodontal surgical procedures at the involved sites.
* Pregnant and lactating women.
* Patients on medications known to interfere with periodontal tissue health or healing.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-01 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Percentage of Mean Root Coverage | 6 months
Complete Root Coverage | 6 months
Root Coverage Esthetic Score | 6 months
Recession Depth Reduction | 6 months

SECONDARY OUTCOMES:
Gingival Recession Width Reduction | 6 months
Probing Depth (PD) | 6 months
Clinical Attachment Level (CAL) | 6 months
Keratinized Tissue Width (KTW) | 6 months
Bleeding Index (BI) | 6 months
Gingival Index (GI) | 6 month
Plaque Index | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Joann P George, MDS, Study Director — Krishnadevaraya College of Dental Sciences and Hospital, Krishnadevarayanagara, Hunsamaranahalli, International Airport Road, Bangalore 562157
Locations (1):
- Krishnadevaraya College of Dental Sciences and Hospital, Bangalore, Karnataka, India